CLINICAL TRIAL: NCT02923947
Title: Open-label,Non-randomised,Multicentre,Phase I Study to Assess the Pharmacokinetics, Safety & Tolerability of Osimertinib Following a Single Oral 80mg Dose to Patients w/ Adv Solid Tumours & Normal Renal Function or Severe Renal Impairment.
Brief Title: Study to Assess Osimertinib in Patients w/ Adv Solid Tumours & Normal Kidney Function or Severe Kidney Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00035
Record Dates: First submitted 2016-09-13; First posted 2016-10-05 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumours
Keywords: Pharmacokinetics,; Renal impairment,; Safety assessments,; Solid tumours,; EGFRm+; EGFRm+/T790M+ inhibitor
MeSH Terms: conditions — Renal Insufficiency | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal renal function (Experimental): For inclusion in the study as a patient with normal renal function, patients must have creatinine clearance ≥90 mL/min.
  Interventions: Drug: Osimertinib; AZD9291
- Severe renal impairment (Experimental): For inclusion in the study as a patient with severe renal impairment, patients must have stable severe renal impairment (creatinine clearance <30 mL/min), as defined by the Cockcroft Gault equation, for at least 2 months prior to Day 1.
  Interventions: Drug: Osimertinib; AZD9291

INTERVENTIONS:
Drug: Osimertinib; AZD9291 — 80mg tablet dose to be taken orally - single dose in part A, daily dosing in Part B and continued access until progression or no longer receiving benefit
  Other Names: TAGRISSO™

SUMMARY:
The purpose of this study is to assess the effect of severe renal impairment on the levels of AZD9291 in the blood in patients with advanced solid tumours compared to patients with normal renal function

DETAILED DESCRIPTION:
This is a 3-part study (Part A, Part B and continued access) in patients with advanced solid tumours (excluding lymphoma) that are refractory to standard therapies or for which no standard therapies exist.

Part A will have a non-randomised, open-label, parallel group, multi-centre design to investigate the pharmacokinetics (PK) of a single dose of osimertinib in patients with severe renal impairment compared with patients with normal renal function. Patients with severe renal impairment will be recruited before those with normal renal function to allow the cohorts to be matched as closely as possible in terms of demographic characteristics (ie, age, body mass index [BMI] and sex).

Approximately 16 patients (8 with severe renal impairment and 8 with normal renal function) are planned to be enrolled to obtain at least 12 evaluable patients (6 with severe renal impairment and 6 with normal renal function) in Part A. A patient with severe renal impairment (as measured by the Cockcroft-Gault equation) is defined as having a creatinine clearance (CrCl) of <30 mL/min whilst a patient with normal renal function has a CrCl of ≥90 mL/min. Both the severe renal impairment and normal renal function patients will be recruited such that both groups will be matched for age, sex, and BMI to the maximum extent possible.

In Part A, each patient will receive a single oral dose of osimertinib 80 mg (given as a tablet). Where possible, patients will check into the clinic on Day -1, the evening prior to dosing (Day 1), and remain resident until 24 hours after the dose of osimertinib (Day 2) for collection of blood samples and 24-hour pooled urine for PK analysis during this time. Samples will be analysed to determine the concentrations of osimertinib and metabolites (AZ5104 and AZ7550) in plasma, urine, and plasma ultrafiltrate (PUF). Patients will then return to the clinic as outpatients for assessments on Day 3 (48 hours), Day 4 (72 hours), Day 6 (120 hours), Day 8 (168 hours) and Day 10 (216 hours).

Part B will allow patients with severe renal impairment, who complete Part A, to continue to receive osimertinib 80 mg once daily for 12 weeks and will provide additional safety data. Patients should start Part B after the last PK sample collected in Part A (ie, 216 hours after receiving the single dose of osimertinib in Part A).

If a patient does not immediately continue into Part B, this should be discussed on a case by case basis with the AstraZeneca physician or representative. Patients who enter Part B, will have weekly clinic visits for the first 3 weeks; thereafter visits will be every 3 weeks until Week 12. Safety assessments will be collected and there will be no formal evaluation of efficacy.

At the end of Part B, those patients with severe renal impairment who are deemed to be gaining clinical benefit from osimertinib will enter the continued access phase. Patients with normal renal function can enter the continued access phase immediately after completing Part A (ie, collection of the last PK sample scheduled on Day 10 of Part A). During the continued access phase, patients may continue to take osimertinib 80 mg once daily, if patients and the Investigator deem it appropriate, or until such time as their disease progresses, the Investigator believes the patients are no longer deriving clinical benefit, or patients stop taking osimertinib for any other reason. No clinical data, other than serious adverse events (SAEs) that may be related to the investigational product (IP), will be collected during this phase.

ELIGIBILITY:
Inclusion criteria:

1. For inclusion as a patient with severe renal impairment patient must have stable severe renal impairment (CrCl <30 mL/min at screening), for at least 2 months prior to the study.
2. For inclusion as a patient with normal renal function, patient must have CrCl ≥90 mL/min at screening.
3. >18 years old
4. Histological or cytological confirmation of a solid, malignant tumour (excluding lymphoma) that is refractory to standard therapies or for which no standard therapies exist. Tumours in which inhibition of the EGFR pathway is considered relevant by the Investigator are not mandated but are encouraged.
5. ECOG performance status ≤2
6. Life expectancy of ≥12 weeks
7. BMI 18-35.
8. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to dosing if of child-bearing potential or must have evidence of non-child bearing potential
9. Males should use barrier contraception until 6 months after the last study drug is taken.

Exclusion criteria

1. Participation in another clinical study with an IP during the last 14 days (or a longer period, depending on the agents used).
2. Treatment with any of the following:

   * Treatment with a 1st or 2nd generation EGFR-TKI within 8 days or approximately 5 half-lives, prior to the first dose of study drug.
   * Any cytotoxic chemotherapy, investigational agents or anticancer drugs within 14 days of the first dose of study drug.
   * Osimertinib in the present study or has previously received a 3rd generation EGFR-TKI (eg, CO 1686).
   * Major surgery within 4 weeks of the first dose of study drug.
   * Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment
   * Currently receiving medications or herbal supplements known to be potent inducers of CYP3A4. Patients in Part B and continued access must avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known potent inducer effects on CYP3A4.
3. Patients with severe renal impairment only: use of concurrent medication known to affect CrCl within 7 days of the first dose
4. Unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment; with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy
5. Spinal cord compression or brain metastases, unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment
6. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count <1.5 x 109/L
   * Platelet count <100 x 109/L
   * Haemoglobin <90 g/L
   * ALT >2.5 times the ULN if no demonstrable liver metastases or >5xULN in the presence of liver metastases
   * AST >2.5xULN if no demonstrable liver metastases or > 5xULN in the presence of liver metastases
   * Total bilirubin >1.5 times ULN if no liver metastases or >3xULN in the presence of liver metastases
7. Any of the following cardiac criteria:

   * Mean resting QT interval QTcF >470 msec, obtained from 3 ECGs.
   * Abnormalities in rhythm, conduction or morphology of resting ECG
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
8. Unable to swallow oral medication or patients with GI disorders or significant GI resection.
9. Medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
10. Severe portal hypertension or surgical porto-systemic shunts.
11. Kidney transplant
12. On dialysis

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to infinity for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs post-dose
  Part A: To investigate the PK of osimertinib after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Maximum plasma concentration for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs post-dose
  Part A: To investigate the PK of osimertinib after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero to the last quantifiable time point for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Area under the plasma concentration-time curve from zero to 24 hours post-dose for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Time to maximum plasma concentration for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Apparent clearance following oral administration for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Apparent volume of distribution for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Terminal rate constant for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Terminal half-life for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Amount excreted in urine from time zero to 24 hours post-dose for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Renal clearance for osimertinib | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24hrs post-dose for osimertinib plasma and 24 hour urine collection.
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Maximum plasma concentration for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Maximum plasma concentration for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Time to maximum plasma concentration for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Time to maximum plasma concentration for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Area under the plasma concentration time curve from zero to infinity for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Area under the plasma concentration time curve from zero to infinity for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Area under the plasma concentration-time curve from zero to the last quantifiable time point for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Area under the plasma concentration-time curve from zero to the last quantifiable time point for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Amount excreted in urine from time zero to 24 hours post-dose for AZ5104 | 24 hour pooled collection starting from time of dosing on Day 1
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Amount excreted in urine from time zero to 24 hours post-dose for AZ7550 | 24 hour pooled collection starting from time of dosing on Day 1
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Terminal rate constant for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Terminal rate constant for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Terminal half-life for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Terminal half-life for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Renal clearance for AZ5104 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24hrs post-dose for AZ5104 plasma and 24 hour urine collection.
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Renal clearance for AZ7550 | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24 hours post-dose for AZ7550 plasma and 24 hour urine collection.
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Metabolite to parent ratios for maximum plasma concentration | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Metabolite to parent ratios for area under the plasma concentration time curve from zero to infinity | On Day of dosing in Part A - predose, 1, 2, 4, 6, 8, 10, 24, 48, 72, 120, 168, 216hrs for osimertinib post-dose
  Part A: To investigate the PK of osimertinib and metabolites (AZ5104 and AZ7550) after a single oral dose of 80 mg in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part A: Adverse Events's, graded by the National Cancer Institute Common Terminology Criteria for Adverse Event's (CTCAE v4.0) | Until 30 days following the final dose of osimertinib
  Part A: To investigate the safety and tolerability of a single oral dose of osimertinib in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part A: physical exam | Until 30 days following the final dose of osimertinib
  Part A: To investigate the safety and tolerability of a single oral dose of osimertinib in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part A: vital signs | Until 30 days following the final dose of osimertinib
  Part A: To investigate the safety and tolerability of a single oral dose of osimertinib in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part A: ECG | Until 30 days following the final dose of osimertinib
  Part A: To investigate the safety and tolerability of a single oral dose of osimertinib in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part A: evaluation of laboratory | Until 30 days following the final dose of osimertinib
  Part A: To investigate the safety and tolerability of a single oral dose of osimertinib in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part A: echocardiogram/MUGA. | Until 30 days following the final dose of osimertinib
  Part A: To investigate the safety and tolerability of a single oral dose of osimertinib in patients with advanced solid tumours and normal renal function or severe renal impairment.
Part B - Adverse events, graded CTCAE v4.0 | Until 30 days following the final dose of osimertinib
  Part B: To investigate the safety and tolerability of multiple oral doses of osimertinib in patients with advanced solid tumours and severe renal impairment.
Part B -physical exam | Until 30 days following the final dose of osimertinib
  Part B: To investigate the safety and tolerability of multiple oral doses of osimertinib in patients with advanced solid tumours and severe renal impairment.
Part B - vital signs | Until 30 days following the final dose of osimertinib
  Part B: To investigate the safety and tolerability of multiple oral doses of osimertinib in patients with advanced solid tumours and severe renal impairment.
Part B - ECG | Until 30 days following the final dose of osimertinib
  Part B: To investigate the safety and tolerability of multiple oral doses of osimertinib in patients with advanced solid tumours and severe renal impairment.
Part B - evaluation of laboratory parameters. | Until 30 days following the final dose of osimertinib
  Part B: To investigate the safety and tolerability of multiple oral doses of osimertinib in patients with advanced solid tumours and severe renal impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ravaud, MD, Principal Investigator — Columbia University
Locations (8):
- France (5):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Saint-Herblain
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Madrid
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Vishwanathan K, Sanchez-Simon I, Keam B, Penel N, de Miguel-Luken M, Weilert D, Mills A, Marotti M, Johnson M, Ravaud A. A multicenter, phase I, pharmacokinetic study of osimertinib in cancer patients with normal renal function or severe renal impairment. Pharmacol Res Perspect. 2020 Aug;8(4):e00613. doi: 10.1002/prp2.613. PMID 32567817